CLINICAL TRIAL: NCT04520516
Title: Trial of Auricular Vagus Nerve Stimulation in Painful and Inflammatory Erosive Hand Osteoarthritis
Brief Title: Auricular Vagus Nerve Stimulation in Painful and Inflammatory Erosive Hand Osteoarthritis
Acronym: ESTIVAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Schwa medico (device lending) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: APHP200014
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis; Musculoskeletal Pain; Erosive Osteoarthritis
Keywords: Musculoskeletal pain; Osteoarthritis; Neuromodulation
MeSH Terms: conditions — Osteoarthritis; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tVNS active device (Experimental): VAGUSTIM device from Schwa-Medico Length of use : 12 weeks
  Interventions: Device: Active VAGUSTIM device
- Sham tVNS device (Sham Comparator): Sham VAGUSTIM device from Schwa-Medico Length of use : 12 weeks
  Interventions: Device: Sham VAGUSTIM device

INTERVENTIONS:
Device: Active VAGUSTIM device — Settings: 25 Hz stimulation, 100 microsec pulse width, intensity escalation up to 8 mA or below if tingling sensation, 20 min/day of stimulation in one daily session
  Arms: tVNS active device
Device: Sham VAGUSTIM device — The sham device : no electrical signal for VNS will be delivered.
  Arms: Sham tVNS device

SUMMARY:
Erosive hand osteoarthritis (EHOA) is a difficult-to-treat subtype of HOA characterized by local and systemic low-grade inflammation as well as by high level of pain and of disability.

Auricular transcutaneous vagus nerve stimulation (tVNS) is a promising therapeutic strategy that may reduce inflammation and pain level.

ESTIVAL is a 12 weeks randomized sham-controlled trial investigating the symptomatic efficacy and safety of tVNS in patients with symptomatic and inflammatory EHOA.

tVNS will be performed using a transcutaneous electrical nerve stimulation (TENS) device connected to an auricular electrode stimulating the cutaneous area of the left ear innervated by the auricular ascendant branch of the vagus nerve.

The active and sham device's will display similar appearance but the sham one will not give electric signal.

DETAILED DESCRIPTION:
Symptomatic hand osteoarthritis (HOA) affects 8-16% of the general population above 50 years and involves interphalangeal (IP) joints. HOA symptoms include pain, stiffness and are responsible for disability and substantial burden. Erosive HOA (EHOA) (10% prevalence among symptomatic HOA from the general population and 40-50% prevalence in tertiary centers) is the most severe HOA phenotype characterized by inflammatory flares, more IP joint destruction, pain, soft swelling joints (ie, synovitis), and more disability (similar to rheumatoid arthritis (RA)) than its non-erosive counterpart.

Current symptomatic pharmacological treatments of HOA or EHOA have a poor efficacy on pain (ie, paracetamol) or safety issues (ie, non-steroidal anti-inflammatory drugs (NSAIDs)) in this aging population with frequent comorbidities. Systemic and joint inflammation contribute to EHOA but 4 studies using TNF inhibitors, 2 using hydroxychloroquine, 1 using methotrexate and 1 using a new anti-IL1α/β failed to show any efficacy on pain in HOA or in EHOA. Therefore, innovative therapeutic approaches are awaited.

Stimulation of the vagus nerve (VNS), belonging to parasympathetic system, dampens pro-inflammatory cytokines production by splenic macrophages, through to the binding of acetylcholine neurotransmitter to α7nicotinic receptor on macrophages: this is the cholinergic anti-inflammatory pathway (CAP). VN stimulation (VNS) by cervical implantable device activating CAP has given promising results in refractory RA patients. Beyond its anti-inflammatory effects, VNS is analgesic in chronic pain disorders (headache, fibromyalgia). However, the use of such implantable device is limited by the need of cervical surgery and subsequent potential side effects.

Besides implantable devices, VNS may be also performed using transcutaneous VNS (tVNS) of the ascendant auricular branch of the VN that selectively innervates the cutaneous zone of cymba conchae at the left ear. Auricular tVNS avoids invasive neurosurgery and its potential side effects and is less expensive than implantable VNS, making it an attractive candidate for neurostimulation. Auricular tVNS has given positive results in chronic migraine and is currently tested in RA, Crohn's disease, widespread pain, irritable bowel syndrome and musculoskeletal pain related to systemic lupus.

We hypothesize that auricular tVNS using a transcutaneous electrical nerve stimulation (TENS) device could be a novel, simple and well-tolerated analgesic and anti-inflammatory treatment of symptomatic (i.e., painful) and inflammatory EHOA.

ESTIVAL is a 12 weeks randomized sham-controlled trial investigating the symptomatic efficacy and the safety of tVNS in patients with symptomatic and inflammatory EHOA.

tVNS will be performed using an active or sham transcutaneous electrical nerve stimulation (TENS) device connected to an auricular electrode stimulating the cutaneous area of the left ear innervated by the auricular ascendant branch of the vagus nerve.

Exploratory and ancillary studies will include i) changes of serum biomarkers of inflammation and of cartilage degradation that will be assess at inclusion and at week 12 ii) hand MRI at W0 and W12 of the most symptomatic joint at inclusion for HOAMRIS socring at W0 and W12 for the center of Saint Antoine.

A phone call at D7± 3 days by the clinical research technician or the clinical nurse or the doctor who has performed the education during the D0 visit to check the proper use of the device.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptomatic HOA according to the American College of Rheumatology criteria
* Erosive HOA according to hand radiographs performed in routine practice showing ≥1 erosive digital joint based on Verbruggen-Veys scoring definition
* Hand pain level ≥ 40/100 mm on VAS at inclusion at least half of days of the 30 last days
* At least ≥1 symptomatic IP joint with clinical soft swelling or erythema at inclusion
* reported inadequate response or adverse effects or contraindication with existing medication (including acetaminophen, oral NSAIDs)
* Informed written consent
* Patient affiliated to a social security scheme NB: Clinical inflammation, ultrasound abnormalities and radiographic erosions have not have to be present in the same joint.

Exclusion Criteria:

* Isolated thumb-base OA (i.e., rhizarthrosis)
* Predominance of the pain in the thumb base rather than digital pain
* Other inflammatory joint disease (e.g. gout, reactive arthritis, rheumatoid arthritis, psoriatic arthritis, Lyme disease)
* Psoriasis
* Current skin disease of the left ear (e.g., eczema, urticarial lesion, skin infection, external otitis)
* Ear canal not adapted to apply the auricular electrode
* Known history of cardiac rhythm disturbances, atrio-ventricular block > first degree, or total bundle branch block
* Symptomatic orthostatic hypotension or repeated vasovagal syncope history
* History of vagotomy
* Severe Asthma
* Treated sleep apnea
* Existence of a pain syndrome of the upper limbs, which would interfere with the monitoring of pain
* Fibromyalgia
* Use of other electrically active medical devices (e.g. pacemaker, TENS for chronic pain)
* Use of oral, intramuscular or intra-articular or intravenous steroids, other anti-synovial agents (e.g. slow-acting anti-rheumatic drugs such as methotrexate, sulfasalazine), intra-articular hyaluronic acid to the hand joints within the last 3 months
* Any new hand OA treatment in the previous 2 months, including physiotherapy and provision of new hand splint.
* Planned hand surgery in the next 3 months.
* Use of any investigational (unlicensed) drug within 3 months prior to screening.
* Evidence of serious uncontrolled concomitant medical condition, including cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, gastro-intestinal disease or epilepsy, which in the opinion of the investigator makes them unsuitable for the study
* Pregnant or breastfeeding woman
* Patient under legal protection measure (tutorship or curatorship) and patient deprived of freedom
* Use of VNS before the study
* Use of NSAIDs or paracetamol less than 48h before the D0 visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Day 0 to Week 12 of self-reported hand pain | 12 weeks
  Change from Day 0 to Week 12 of self-reported hand pain in the previous 48 hours measured on a 100 mm visual analogue scale (VAS) : "How much pain in your hands did you experience during the past 48 h?"

SECONDARY OUTCOMES:
AUStralian CANadian Osteoarthritis Hand Index (AUSCAN)(pain, function, stiffness). | Between week 0 and week 12
  AUStralian CANadian Osteoarthritis Hand Index (AUSCAN) 3.1 pain, function and stiffness subscores (for each subscore: 0-100 mm scale)
Modified Functional Index for Hand OsteoArthritis (FIHOA) | Between week 0 and week 12 vvv
  scale minimum 0 , and maximum 30.
Cochin Hand Function Scale. | Between week 0 and week 12
Percentage of patients below the Patient Acceptable Symptom State (PASS) of pain (VAS<40/100) | Between week 0 and week 12
EuroQoL EQ-5D. | Between week 0 and week 12
Hospital Anxiety and Depression Scale (HAD). | Between week 0 and week 12 vvvvvvv
Fatigue intensity on a 0-100 mm VAS | Between week 0 and week 12
Number of painful hand joints (0-30) under pressure. | Between week 0 and week 12
Number of swollen hand joints (0-30). | Between week 0 and week 12
Patient Global Assessment (PGA) of health status on a 0-100 mm VAS. | Between week 0 and week 12
DN-4 Questionnaire evaluating neuropathic pain. | Between week 0 and week 12
Change over time of VAS pain. | Week 0, Week 4, Week 8, and Week 12
Change over time of FIHOA. | Week 0, Week 4, Week 8, and Week 12
Change over time of AUSCAN (pain, stiffness, and function). | Week 0, Week 4, Week 8, and Week 12
Percentage of patients with symptom levels below which they consider their condition acceptable (PASS), defined by a VAS <40/100 | Week 12
Proportion of OMERACT-OARSI responders. | Week 12
Percentage of responders according to the Patient Global Impression of Change (PGIC) score | Week 12
Total paracetamol consumption (g) divided by treatment duration using a patient-filled diary. | Between week 0 and week 12
Change in percentage in serum inflammatory or pain-related markers | Between week 0 and week 12
Change in serum cartilage degradation markers (Coll2-1 (a marker of type II collagen denaturation), Coll2-1-NO2). | Between week 0 and week 12
Proportion of side effects | 4 weeks, 8 weeks and 12 weeks
  report of side effects during the study period
Average daily use duration and cumulative use duration of the Vagustim device since the last visit, collected from the device's tracking system before each visit. | Between week 0 and week 12

OTHER OUTCOMES:
W0-W12 change in the WOMAC for other osteoarthritis sites (hips, knees) if present at inclusion. | Between week 0 and week 12
Effectiveness of the blinding procedure and the ease of use of the device | Week 12
  * Patient satisfaction with the treatment, assessed on a 5-point scale (from very satisfied to not at all satisfied).
  * Ease of use assessed on a 4-point scale (from very easy to very difficult).
  * Indication by patients whether they believe they received the active or sham device. d. Indication by the investigator whether they believe the patient received the active or sham device.
Change in HOAMRIS subscores of synovitis and subchondral bone marrow edema using MRI examination | Between week 0 and week 12
Clinical efficacy (primary endpoint and the OMERACT-OARSI response) according clinical, biological or radiographic characteristics at inclusion | Between week 0 and week 12
Correlation between baseline biological biomarkers and clinical response in the active group | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie SELLAM, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Rhumatologie - Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Courties A, Tuffet S, Cormier G, Roux CH, Ornetti P, Pers YM, Gottenberg JE, Lespessailles E, Chapurlat R, Arniaud D, Rannou F, Wendling D, Eymard F, Mathieu S, Richette P, Saraux A, Marotte H, Poursac N, Rat AC, Bastard JP, Fellahi S, Henrotin Y, Minssen L, Deprouw C, Nguyen C, Touati A, Berard L, Rousseau A, Simon T, Maheu E, Berenbaum F, Sellam J. Transcutaneous auricular vagus nerve stimulation versus sham stimulation in patients with erosive hand osteoarthritis (ESTIVAL): a randomised, multicentre, double-blind, sham-controlled trial. Lancet Rheumatol. 2026 Feb;8(2):e98-e107. doi: 10.1016/S2665-9913(25)00226-7. Epub 2025 Dec 8. PMID 41380709
- [Derived] Courties A, Deprouw C, Rousseau A, Berard L, Touati A, Kalsch J, Villevieille M, Maheu E, Miquel A, Simon T, Berenbaum F, Sellam J; ESTIVAL study group. Transcutaneous vagus nerve stimulation in erosive hand osteoarthritis: protocol for the randomised, double-blind, sham-controlled ESTIVAL trial. BMJ Open. 2022 Mar 22;12(3):e056169. doi: 10.1136/bmjopen-2021-056169. PMID 35318234